CLINICAL TRIAL: NCT06927232
Title: Azacitidine Plus Luspatercept Versus Azacitidine Monotherapy in Higher-risk Myelodysplastic Neoplasms: a Randomized Prospective Study
Brief Title: AZA+Lus VS AZA Monotherapy in HR-MDS
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Bing Han, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AZA-Lus-HRMDS
Record Dates: First submitted 2025-04-01; First posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Higher-risk Myelodysplastic Syndrome
Keywords: luspatercept; azacitidine; higher-risk myelodysplastic syndrome
MeSH Terms: interventions — Azacitidine; luspatercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Azacitidine+Luspatercept (Experimental)
  Interventions: Drug: Azacitidine (AZA); Drug: Luspatercept
- Azacitidine (Active Comparator)
  Interventions: Drug: Azacitidine (AZA)

INTERVENTIONS:
Drug: Azacitidine (AZA) — Azacitidine 75mg/m/ day *5 days, 28 days for 1 course
Drug: Luspatercept — Luspatercept 1.0 mg/kg subcutaneously every 3 weeks, adjusted according to hemoglobin, up to 1.75mg/kg. If hemoglobin ≥120g/L, luspatercept can be discontinued.
  Arms: Azacitidine+Luspatercept

SUMMARY:
This study is a randomized, prospective, single-center, open-label cohort study involving untreated HR-MDS patients. The patients were divided randomized into AZA+Lus cohort and AZA monotherapy cohort.

DETAILED DESCRIPTION:
The hypomethylating agents (HMA) azacitidine (AZA) and decitabine (DEC) have been shown to improve survival and delay disease progression in patients with high-risk MDS. They are recommended by the NCCN as first-line treatments for patients with high-risk MDS. Clinical trials have demonstrated an OR rate of approximately 40-50% with AZA in patients with high-risk MDS. Despite the efficacy of HMA therapy, the rate of transfusion independence remains low. Anemia remains the most prominent symptom in refractory patients, with very limited options for subsequent treatment. Prolonged anemia affects every organ function and seriously affects the prognosis of patients.

Luspatercept is currently approved for the treatment of patients with both erythropoiesis receptor agonist ( ESA) treatment failures in transfusion-dependent low-risk MDS-RS patients. In a randomized controlled phase III clinical trial, compared to a placebo group, luspatercept significantly improved transfusion dependence and improved hemoglobin and quality of life in refractory MDS-RS patients. A recent conference report suggested that there was no significant difference in efficacy between low-risk and high-risk patients treated with luspatercept and that the HI rate for high-risk patients treated with luspatercept monotherapy was approximately 50%.

Thus this study aimed to compare the efficacy of AZA+luspatercept and AZA monotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* Diagnosed as higher-risk MDS (IPSS intermediate-2/high-risk, or IPSS-R >3.5, or IPSS-M moderate high-, high-, very high-risk)
* Untreated patients
* Liver and kidney function less than 2 times of upper limit of normal
* ECOG≤2 and expected survival more than 6 months
* Informed consent signed

Exclusion Criteria:

* With active infection
* Other malignant tumors
* Obvious abnormal liver and kidney function, or abnormal function of other organs
* Combined with myelofibrosis
* Have undergone bone marrow transplantation
* Pregnant or lactating women, or men who have recent reproductive needs
* Allergic to azacytidine, Rotercept or excipients
* History of polysorbate 80 allergy
* Refuse to sign informed consent
* Researchers consider it inappropriate to participate in the experiment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | 3 months, 6 months

SECONDARY OUTCOMES:
complete response rate | 3 months, 6 months
rate of transfusion independence | 3 months, 6 months
adverse event rate | through study completion, an average of 1 year
relapse rate | through study completion, an average of 1 year
progress-free survival | through study completion, an average of 1 year
overall survival | through study completion, an average of 1 year